CLINICAL TRIAL: NCT03932175
Title: Effects of a Behavioural Intervention in Home-based Mechanically Ventilated Patients
Brief Title: Behavioural Intervention in Mechanically Ventilated Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, CRISTINA EMBID LOPEZ, Doctor, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NIV - MyPathway
Record Dates: First submitted 2019-04-26; First posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Noninvasive Ventilation; Chronic Disease Lung

STUDY DESIGN:
Intervention Model Description: Two-groups, randomised parallel study with 1:1 ratio
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will assess only anonymized data from the two study groups, wherein every group will also be de-identified in relation to its study arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The multicomponent intervention will comprise three aspects on-top of usual care: i) Motivational interview to assess patient's adherence profile and to raise the compromise with the behaviour change towards NIV, physical activity and nutritional habits; ii) Bi-directional interaction between the study participants and clinical staff delivered by the MyPathway app, where specific clinical problems regarding NIV will be addressed as they arise; and iii) Motivational messages and educational material delivered via the MyPathway app regarding changes in physical activity and/or nutritional habits. As part of the behavioural intervention, goal setting for NIV adherence and life-style changes will be introduced to the MyPathway app in order for the participants to follow the advice.
  Interventions: Behavioral: Intervention group
- Control group (No Intervention): Patients will receive usual care according to guidelines on management of chronically ventilated patients, without any mHealth tool or behavioural intervention

INTERVENTIONS:
Behavioral: Intervention group — Behaviorial intervention on non-invasive ventilation use and adherence alongside lifestyle changes recommendations supported by an mHealth tool (MyPathway app)
  Arms: Intervention group

SUMMARY:
Background: Non-invasive ventilation at home for chronic respiratory failure due to different etiologies has proven effective regarding mortality and quality of life. Nonetheless, adherence to therapy still constitutes a clinical day-to-day problem. Physiological monitoring has shown to improve adherence. We hypothesise that an additional behavioural intervention delivered via mHealth tools, on top of usual care, can further enhance therapeutical success alongside patient satisfaction.

Methods: Randomized single-blinded controlled trial with an intervention and control groups. Intervention will consist of a multi-component based behavioural intervention delivered via a mHealth tool, during a three-month period. Primary objective will be change in self-efficacy towards non-invasive ventilation use

Statistical Analysis: Based on a change of 0.5 units in the Self Efficacy in Sleep apnea (SEMSA) questionnaire, a sample size of 30 subjects per study arm was calculated. It has been anticipated a drop-out rate of 5%. Standard statistical analysis will take place.

Expected results: we expect a positive change on the SEMSA score (reflecting better self-efficacy) after three-month use. Indirectly, this enhancement should facilitate patient adherence specifically via mask leak problems resolution. Also, we presume that the proposed mHealth tool will be highly usable and accepted by the patients, leading to overall satisfaction with the service provided.

DETAILED DESCRIPTION:
The polio epidemics demonstrated the safety and efficacy of non-invasive ventilation (NIV) to decrease mortality. Since then, this therapeutic approach has been shown to reduce hospital admissions, impact favourably on health-related quality of life (HRQL), improve sleep quality and reduce mortality in patients with diverse chronic pathologies. This success has driven the increase in prevalence of patients using home NIV in Europe, ranging from 4.5 to 20 per 100,000 adults.

The use of NIV at home has been proven to be cost-effective, but patients' adherence to therapy has still potential to improve which should further enhance healthcare efficiencies of the intervention. Optimization of physiological settings and monitoring can contribute to enhance adherence by improving timely detection of problems such as mask leaks, patient-ventilator asynchronies, etc. However, improvement of behavioural aspects such as patient motivation and empowerment for self-management are also important factors to consider when addressing adherence to respiratory therapies.

The current protocol seeks to explore the transfer of previous positive experiences on behavioural interventions in other fields (i.e. physical activity into home-based NIV and, in general, into respiratory therapies. Specifically, we will explore the concept of self-efficacy. It is defined as the individual's perceived capability to perform the particular behaviour. A person who does not believe in her or his own capability to perform a desired action will fail to adopt, initiate, and maintain it. Self-efficacy is therefore seen as the most influential motivational factor and the strongest predictor of behavioural intentions.

The application of self-efficacy to the problem of identifying predictors of BIPAP use derives from the social cognitive theory concept of Bandura (Bandura's model). This model has been widely applied in studies of the adoption, initiation, and maintenance of health-promoting behaviors and consists of the concepts of perception of the risk to health, expectations regarding treatment outcome (outcome expectancies), and the confidence or volition to engage in the behavior (treatment self-efficacy).

Alongside this well-defined behavioural concept, we also identify the role of information and communication technologies (ICT) as a promising scenario to generate efficiencies by enhancing coordination between stakeholders and contributing to improve health outcomes.

Nonetheless, it is acknowledged that the scenario is not still mature. Mainly, because of lacking evidence in real-world scenarios for the capacity of ICT to escort behavioural changes in chronic complex patients. It is widely accepted that, despite current limitations, chronic complex patients are an ideal population where care coordination, patient and medical staff satisfaction alongside patient empowerment are of utmost importance to produce health benefits.

The study protocol intends to produce evidence on the capacity of a behavioural intervention to increase patient empowerment for self-management and adherence to therapy accompanied by an ICT tool interoperable with the information system of the healthcare provider. Moreover, the intervention should generate high acceptability/satisfaction among patients, carers and professionals. We fully acknowledge that if the expected results are achieved, the proposed study shall be followed by long-term assessment of the impact of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients with hypercapnic ventilatory failure due to chest wall, neuromuscular, lung parenchyma and/ or airway disease already receiving treatment with non-invasive ventilation irrespective of treatment duration.
* Having a mobile phone, tablet or personal computer that can support the use of MyPathway application.
* Accepting to participate in the study and signing informed consent.

Exclusion Criteria:

* Clinical instability (including a respiratory acute exacerbation) at time of assessment for study enrolment.
* Not willing to use the proposed mHealth tool at home.
* Severe psychiatric disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-06-19 (Estimated); Study Completion 2019-06-25 (Estimated)

PRIMARY OUTCOMES:
Self efficacy | 3 months
  Change in the Self Efficacy in Sleep apnea (SEMSA) questionnaire

SECONDARY OUTCOMES:
mHealth tool usability | 3 months
  mHealth tool usability assessed by the System Usability Scale
Patient satisfaction | 3 months
  Patient satisfaction with the mHealth tool assessed by the Net Promoter Score
Non-invasive ventilation adherence | 3 months
  Number of hours of daily use of the non-invasive ventilation machine during the study period
Patient centred healthcare provision | 3 months
  Patient centred healthcare provision as measured by the Person Centred Coordinated Experience Questionnaire
Continuity of care within the healthcare system | 3 months
  Continuity of care within the healthcare system as measured by the Nijmegen Continuity of Care Questionnaire
Health and well-being | 3 months
  Change in quality of life assessed by the EuroQol-5D questionnaire
Sleepiness | 3 months
  Change in sleepiness assessed by the Epworth Sleepiness Score

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Embid, MD, Principal Investigator — Hospital Clinic
Locations (1):
- Hospital Clinic, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lloyd-Owen SJ, Donaldson GC, Ambrosino N, Escarabill J, Farre R, Fauroux B, Robert D, Schoenhofer B, Simonds AK, Wedzicha JA. Patterns of home mechanical ventilation use in Europe: results from the Eurovent survey. Eur Respir J. 2005 Jun;25(6):1025-31. doi: 10.1183/09031936.05.00066704. PMID 15929957
- [Background] de Lucas Ramos P, Rodriguez Gonzalez-Moro JM, Paz Gonzalez L, Santa-Cruz Siminiani A, Cubillo Marcos JM. [Current status of home mechanical ventilation in Spain: results of a national survey]. Arch Bronconeumol. 2000 Nov;36(10):545-50. Spanish. PMID 11149196
- [Background] Barberan-Garcia A, Ubre M, Roca J, Lacy AM, Burgos F, Risco R, Momblan D, Balust J, Blanco I, Martinez-Palli G. Personalised Prehabilitation in High-risk Patients Undergoing Elective Major Abdominal Surgery: A Randomized Blinded Controlled Trial. Ann Surg. 2018 Jan;267(1):50-56. doi: 10.1097/SLA.0000000000002293. PMID 28489682
- [Background] Troosters T, Maltais F, Leidy N, Lavoie KL, Sedeno M, Janssens W, Garcia-Aymerich J, Erzen D, De Sousa D, Korducki L, Hamilton A, Bourbeau J. Effect of Bronchodilation, Exercise Training, and Behavior Modification on Symptoms and Physical Activity in Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2018 Oct 15;198(8):1021-1032. doi: 10.1164/rccm.201706-1288OC. PMID 29664681
- [Background] Bandura A. Self-efficacy mechanism in human agency. Am Psychol. 1982;37(2):122-47.
- [Background] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061
- [Background] Ambrosino N, Vitacca M, Dreher M, Isetta V, Montserrat JM, Tonia T, Turchetti G, Winck JC, Burgos F, Kampelmacher M, Vagheggini G; ERS Tele-Monitoring of Ventilator-Dependent Patients Task Force. Tele-monitoring of ventilator-dependent patients: a European Respiratory Society Statement. Eur Respir J. 2016 Sep;48(3):648-63. doi: 10.1183/13993003.01721-2015. Epub 2016 Jul 7. PMID 27390283
- [Derived] Baltaxe E, Embid C, Aumatell E, Martinez M, Barberan-Garcia A, Kelly J, Eaglesham J, Herranz C, Vargiu E, Montserrat JM, Roca J, Cano I. Integrated Care Intervention Supported by a Mobile Health Tool for Patients Using Noninvasive Ventilation at Home: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Apr 13;8(4):e16395. doi: 10.2196/16395. PMID 32281941